CLINICAL TRIAL: NCT01860989
Title: An Open Label, Single Dose Study to Assess Efficacy, Safety, Tolerability and Pharmacokinetics of KAE609 in Adult Patients With Acute, Uncomplicated Plasmodium Falciparum Malaria Mono-infection
Brief Title: A Study to Assess Efficacy, Safety of KAE609 in Adult Patients With Acute Malaria Mono-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKAE609X2202
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Cure Rate
Keywords: parasitemia
MeSH Terms: conditions — Parasitemia | interventions — NITD 609

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 6-12 subjects with Plasmodium falciparum malaria will receive 75 mg KAE609 as a single dose
  Interventions: Drug: KAE609
- Cohort 2 (Experimental): 6-12 subjects with Plasmodium falciparum malaria will receive 150 mg KAE609 as a single dose
  Interventions: Drug: KAE609
- Cohort 3 (Experimental): 6 to 12 subjects with Plasmodium falciparum malaria will receive 225 mg KAE609 as a single dose
  Interventions: Drug: KAE609
- Cohort4 (Experimental): 6- 12 subjects with Plasmodium falciparum malaria will receive 300 mg KAE609 as a single dose
  Interventions: Drug: KAE609

INTERVENTIONS:
Drug: KAE609 — KAE609 75mg single dose
  Arms: Cohort 1
Drug: KAE609 — KAE609 150mg single dose
  Arms: Cohort 2
Drug: KAE609 — KAE609 225mg single dose
  Arms: Cohort 3
Drug: KAE609 — KAE609 300mg single dose
  Arms: Cohort4

SUMMARY:
This study will assess efficacy, safety , tolerability and PK in uncomplicated adult malaria patients with acute P. falciparum infection after single dose with KAE609 at 75 mg, 150mg, 225mg and 300mg/day

DETAILED DESCRIPTION:
the study is comprised of 4 sequential cohorts, in total there will be up to 48 patients enrolled in the study.

cohort 1: 6-12 patients receive 75mg single dose. cohort 2: 6-12 patients receive 150mg single dose. cohort 3: 6-12 patients receive 225mg single dose. cohort 4: 6-12 patients receive 300mg single dose. After approximately every 6 patients in any cohort have been treated with a given dose and complete the first 15 days, a safety and tolerability data review will be conducted by a Data Monitoring Committee(DMC). Consensus agreement of DMC is required to either escalate to the next dose level or expand a given cohort with an additional 6 patients in order to obtain more safety data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 to 60 years
* Presence of mono-infection of P. falciparum
* Weight between 40 kg to 90 kg

Exclusion Criteria:

* Patients with signs and symptoms of severe/complicated malaria
* Mixed Plasmodium infection
* Presence of other serious or chronic clinical condition requiring hospitalization.
* Severe malnutrition
* Significant chronic medical conditions which in the opinion of the investigator preclude enrollment into the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Thailand (3):
  - Novartis Investigative Site, Ratchabari
  - Novartis Investigative Site, Si Sa Ket
  - Novartis Investigative Site, Tak
- Novartis Investigative Site, Hanoi, Vietnam

RESULTS

PARTICIPANT FLOW:
Groups:
- Total - Cohort 1: Cohort 1 6-12 subjects with Plasmodium falciparum malaria will receive 75 mg KAE609 as a single dose
Period: Overall Study
Arm/Group | Total - Cohort 1
Started | 11
Completed | 6
Not Completed | 5
Not completed — Unsatisfactory therapeutic | 5

BASELINE CHARACTERISTICS:
Arm/Group | Total - Cohort 1
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (7.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: 28-day Cure Rate
Description: 28-day cure rate was measured by the endpoint of complete cure without recrudescence before Day 29. The primary variable of 28-day cure rate was defined as the proportion of patients with clearance of asexual parasitemia (by blood film) by day 6 of the study, and without subsequent recrudescence (by blood film).
Time Frame: Day 28
Population: PharmacoDynamic (PD) Analysis Set - All the 11 patients were included in PD analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | Total - Cohort 1
Number analyzed (Participants) | 11
Percentage of participants | 63.67

ADVERSE EVENTS:
Arm/Group | Total - Cohort 1
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total - Cohort 1 (N=11)
Jaundice (Hepatobiliary disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total - Cohort 1 (N=11)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 2
Blood pressure systolic increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Platelet count decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.